CLINICAL TRIAL: NCT03186664
Title: The Role of SAtivex® Associated With Robotic-Rehabilitation in Improving the Motor Performances of Multiple Sclerosis Patients (SARR)
Brief Title: The Role of SAtivex® in Robotic-Rehabilitation
Acronym: SARR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, MD PhD, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/2016
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Rehabilitation
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Sativex+Lokomat Training (Experimental): Patients Sativex responders will perform a neurorobotic-assisted gait training (RAGT, each session will last at least 45', 3 times per week, for a total amount of 20 treatment's sessions).
  Interventions: Device: Lokomat training; Drug: Sativex
- B: other antispastic+Lokomat Training (Active Comparator): Patients treated with others antispastic drugs will perform a neurorobotic-assisted gait training (RAGT, each session will last at least 45', 3 times per week, for a total amount of 20 treatment's sessions).
  Interventions: Device: Lokomat training

INTERVENTIONS:
Device: Lokomat training — The neurorobotic treatment will be performed by using the Lokomat (Lokomat, Hocoma, Volketswil, Switzerland) device. The work load will be progressively adjusted based on the improvement of motor performances. Training parameters (weight support, etc) will be individually adapted. During the first Lokomat session, support will be set at 50% of the body weight and will be adapted on observation of the gait. The Lokomat motor guidance system will be first set at 100%, corresponding to a passive walk.
  Other Names: RAGT
Drug: Sativex — Patients in treatment with Sativex will receive cannabis-based medicine extract presented in a pump action sublingual spray. Sativex is composed of whole cannabis plant extract, containing THC (27 mg/mL) and CBD (25 mg/mL), in ethanol/propylene glycol (50:50) excipient.
  Each actuation delivers 100 KL of spray, containing THC 2.7 mg and CBD 2.5 mg. The number and frequency of dosing (sprays) with Sativex will vary from individual to individual and it may take a number of weeks to find the correct dose of Sativex for the individual patient.
  Other Names: Nabiximols
  Arms: A: Sativex+Lokomat Training

SUMMARY:
Spasticity is frequently experienced by people with Multiple Sclerosis (MS), negatively impacting on patient's motor functional outcome, including walking. Currently, none of the available MS disease-modifying medications has been shown to stop or reverse gait disability. Recently the nabiximols has been tested for the treatment of spasticity and walking impairment in MS. Nabiximols (trade name Sativex®) is an oromucosal spray formulation containing 1:1 fixed ratio of delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) derived from cloned Cannabis sativa L. plant. The main active substance, THC, acts as a partial agonist at human cannabinoid receptors (CB1 and CB2), and may modulate the effects of excitatory (glutamate-GLU-) and inhibitory (gamma-aminobutyric acid -GABA-) neurotransmitters, leading to muscle relaxation, which in turn is responsible for spasticity improvement. Cannabinoid receptors may modulate both excitatory and inhibitory transmission at central synapses, and have been heavily implicated, in animal models, in multiple forms of synaptic plasticity, such as long-term potentiation (LTP) and long-term depression (LTD). Indeed, in a previous study implying transcranial magnetic stimulation (TMS) technique, it has been hypothesized that the activation of cannabinoid receptors by Sativex® could modulate the balance between LTP and LTD like plasticity by changing the state of cortical excitability. In a recently study it has been proposed that Sativex may modulate the cortical excitability changing the activity of inhibitory GABAergic cortico-cortical synapses. Aim of our study is to clarify the role of Sativex coupled to a robotic neurehabilitation training in MS patients in improving the motor outcome, by means of clinical, kinematic, beside some neurophysiological and measures.

DETAILED DESCRIPTION:
Forthy MS patients affected by gait disturbances and moderate-severe spasticity will be enrolled: 20 out of them in treatment with Sativex (Group A) considered as responders and 20 treated only with the most common antispastic used in MS (Group B). All the 40 subjects, divided into two groups (A: Sativex+Lokomat Training and B: other antispastic+Lokomat Training), will perform a neurorobotic-assisted gait training (RAGT, each session will last at least 45', 3 times per week, for a total amount of 20 treatment's sessions). All patients will undergo a complete blind physical and neurological examination, including evaluation of disability by means of the Expanded Disability Scale (EDDS) and assessment of spasticity using the Modified Ashworth Scale (MAS) and the numerical rating scale (NRS). To clarify the role of Sativex® in improving spasticity gait-related symptoms the following scales will be also administered: ten meters walking test (10wt), Ambulation Index (AI). Quality of life will be evaluated by means of MSQOL 54. The skilled clinician will be blind to the drug treatment.Moreover, some electrophysiological parameters to test cortical excitability will be also evaluated: motor evoked potentials (MEP) amplitude, short intracortical inhibition (SICI) and facilitation (ICF) from the abductor pollicis brevis muscle (APB) of the most affected side. The same assessment will be applied in baseline, at the end of the robotic training (T1) and 30 days after the end of the nerehabilitation training (T2).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were:

* age of 18-65 years,
* diagnosis of definite relapsing-remitting or primary-progressive Multiple Sclerosis, -absence of clinical relapses from no gadolinium enhanced lesions on brain and spinal cord MRI performed at least six months prior to study entry,
* no mood or sleep disorders (Hamilton score of <17),
* a moderate to severe spasticity in at least two districts of upper and/or lower limbs; -absence of clinical or neuroradiological relapses from at least six months prior to study entry,
* Expanded Disability Status Scale (EDSS) total score between 3.5 and 7.0,
* no history of psychosis,
* no presence of pace-maker, aneurysms clips, neurostimulator or brain/subdural electrodes (safety TMS procedure),
* right handedness,
* central conduction time in upper limbs of <8 ms;
* no robotic gait traing contraindications.

Exclusion Criteria:

* History of psychosis,
* presence of pace-maker, aneurysms clips, neurostimulator or brain/subdural electrodes (safety TMS procedure),
* central conduction time in upper limbs of <8 ms;
* robotic gait traing contraindications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure | eight months
  Contains 18 items composed of:
  This is divided 13 motor tasks and 5 cognitive tasks, considered basic activities of daily living)
10m walking test | eight months
  A tool to better define gait parameters, with regards to speed.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino-Pulejo", Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No